CLINICAL TRIAL: NCT03066037
Title: Regional-anaesthesiological Infiltration Techniques for the Management of Chronic Pain: a Retrospective Study
Acronym: RetroBlock
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Sascha Tafelski, Physician scientist, Charite University, Berlin, Germany
Other Study IDs: RetroBlock
Record Dates: First submitted 2017-02-20; First posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Chronic Pain; Trigeminal Neuralgia; Cluster Headache; Post-Zoster Neuralgia; Post Zoster Pain; Neuropathic Pain
Keywords: regional-anaesthesiological infiltration; block series; invasive pain treatment
MeSH Terms: conditions — Chronic Pain; Trigeminal Neuralgia; Cluster Headache; Neuralgia, Postherpetic; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: regional-anaesthesiological infiltration — Patients with therapy refractory chronic pain are treated with local infiltration techniques using e.g. local anaesthetics, opioids or drug combinations. Targeted structures are e.g. Ganglion stellatum, Ganglion pterygopallatinum, Trigeminal nerve branches (V1-V3). Patients receive a context- sensitive number of blocks in a series of infiltrations depenting on their pain course.
  Other Names: block series

SUMMARY:
There is a significant debate whether local infiltration techniques may be a method to treat complicated chronic pain syndromes, e.g. refractory headache. Until now there is a lack of evidence regarding efficacy of this treatment especially in long term follow up. Similarly, indication and management are under debate. Aim of this trial is to analyse pain scores during first treatment with anaesthesiological infiltration series.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic pain disease undergoing regional-anaesthesiological infiltration series

Exclusion Criteria:

* pregnancy
* patients in legal custody
* age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are included with any refractory neuropathy, refractory headache or chronic disease with any invasive pain infiltration technique applied. All infiltration series are embedded in multi-modal therapy concepts.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-11-13 (Actual)

PRIMARY OUTCOMES:
NRS reduction during therapy | 2 weeks
  Reduction (relative and absolute) of pain during series of infiltrations comparing NRS scores before and after infiltrations

SECONDARY OUTCOMES:
Number of blocks in a series | 4 weeks
  Number of blocks in a series to achieve the targeted NRS reduction
Time till recurrent pain | 24 weeks
  Time until a new series of blocks is requested by the patient
clinical course of pain | 2 weeks
  NRS development during series of infiltrations
type of infiltration | 2 weeks
  location of infiltrations with medication used
co-parameters of pain chronification | 2 weeks
  co-factors of pain like co-morbidity, duration of pain disease, psychological diseases and association with primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schäfer, Prof., Principal Investigator — Charité University Berlin
Locations (1):
- Charité hospital, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Data sharing can be requested and will be evaluated by Charité data safety authorities.

REFERENCES:
- [Background] Dworkin RH, O'Connor AB, Kent J, Mackey SC, Raja SN, Stacey BR, Levy RM, Backonja M, Baron R, Harke H, Loeser JD, Treede RD, Turk DC, Wells CD. Interventional management of neuropathic pain: NeuPSIG recommendations. Pain. 2013 Nov;154(11):2249-2261. doi: 10.1016/j.pain.2013.06.004. Epub 2013 Jun 6. PMID 23748119
- [Background] Tafelski S, Beutlhauser T, Gouliou-Mayerhauser E, Fritzsche T, Denke C, Schafer M. [Practice of regional anesthesia for chronic pain patients in specialized pain services : A nationwide survey in Germany]. Schmerz. 2015 Apr;29(2):186-94. doi: 10.1007/s00482-014-1503-6. German. PMID 25479710